CLINICAL TRIAL: NCT00791427
Title: ERG/EOG Study in AMD Patients Treated With Ranibizumab
Acronym: FVF4154s
Status: Completed | Type: Observational
Sponsor: Retina Center, Minnesota (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Abdhish R. Bhavsar, M.D., President/Physician/Owner, Retina Center, Minnesota
Other Study IDs: FVF4154s
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- AMD Patients
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — 0.05 ml of ranibizumab injected into the eye monthly for one year

SUMMARY:
This is an open-label study assessing electrophysiologic testing of the retina with Electoretinogram (ERG) /Electrooculogram (EOG) tests in patients with exudative age-related macular degeneration (AMD). The standard FDA-approved treatment for wet AMD is ranibizumab (Lucentis). This study focuses on the ERG and EOG tests to evaluate retinal responses to ranibizumab treatment in AMD.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age >55 years
* Patients to be included in the study must have AMD with choroidal neovascularization
* BCVA between 20/20 - 20/400
* Lesion size less than or equal to 12 MPS disc areas

Exclusion Criteria:

* Prior treatment with an anti-VEGF agent within 6 months of enrollment in this study
* Pregnancy (positive pregnancy test)
* Premenopausal women not using adequate contraception. The following are considered effective means of contraception: surgical sterilization or use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel, an IUD, or contraceptive hormone implant or patch
* Prior enrollment in the study
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
* Participation in another simultaneous medical investigation or trial
* Media insufficient to obtain a view
* Other causes of CNV not related to AMD
* Active ocular or peri-ocular infection
* Ocular surgery within 1 month prior to the study

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will have AMD with choroidal neovascularization and above age 55 years.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2008-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
ERG/EOG | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- The Retina Center, Minneapolis, Minnesota, United States

REFERENCES:
- See also: facility website — http://www.retinadocs.com